CLINICAL TRIAL: NCT04296136
Title: Quality Improvement Project: Assessing the Use of Advanced Care Planning Documentation for Patients at High Risk of 30-day Mortality on Hospital Medicine Services
Brief Title: Quality Improvement Project for Advance Care Planning Tool in Hospital Medicine
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00104527
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Advance Care Planning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High risk of mortality: Adult patients admitted to the hospital medicine service with a high risk of mortality
  Interventions: Other: Advance Care Planning Discussion
- High risk of mortality (pre-implementation): Adult patients admitted to the hospital medicine service with a high risk of mortality

INTERVENTIONS:
Other: Advance Care Planning Discussion — Goals of care discussion with patient, documentation with electronic health record note and advance care planning billing. This will also include: pharmacy review of medications, case management review, and coding specialist review.
  Groups: High risk of mortality

SUMMARY:
Hospitalized patients and their families are often unprepared regarding end-of-life care. Even patients with high risk of mortality within the index admission or 30 days after admission often do not have clearly defined goals of care. This lack of clarity can create difficult scenarios for patients, their families, and care providers. Lack of communication and documentation of these goals can lead to unnecessary tests, procedures, and readmissions. By creating advanced care planning education for the hospital medicine department, a standardized note template, and EMR utilization for storage and reference of patient's goals of care documentation we aim to facilitate the conveyance of patient's wishes/preferences across different care providers and across separate encounters within the healthcare system. For this study, we will use a pre-post study design to evaluate the implementation of this quality improvement intervention.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the inpatient medicine service with high risk of mortality.

Exclusion Criteria:

* Involuntary commitment during the index admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for the QI project will include two groups (pre and post-implementation) in order to evaluate the effectiveness of the program. Both the pre-implementation and the intervention (post-implementation) groups consist of adult patients admitted to the hospital medicine service with a high risk of mortality; clinicians providing care for patients in the post-implementation group will also receive a notification of the patient's high risk of mortality and recommendation for a serious illness conversation. The evaluation has been narrowed to a pre-post study design, which will enable our team to identify the impact of the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 743 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have advanced care planning notes completed during the admission | Hospital admission, up to 7 days
  As measured by medical record review (Pre-implementation)
Proportion of patients who have advanced care planning notes completed during the admission | Hospital admission, up to 7 days
  As measured by medical record review (Post-implementation)

SECONDARY OUTCOMES:
Proportion of patient who have documentation utilizing the electronic health record dotphrase note template | Hospital admission, up to 7 days
  As measured by medical record review (Pre-implementation)
Proportion of patient who have documentation utilizing the electronic health record dotphrase note template | Hospital admission, up to 7 days
  As measured by medical record review (Post-implementation)
Proportion of patients who are billed for advanced care planning | Hospital admission, up to 7 days
  As measured by medical record review (Pre-implementation)
Proportion of patients who are billed for advanced care planning | Hospital admission, up to 7 days
  As measured by medical record review (Post-implementation)
Proportion of patients who receive palliative care consults | Hospital admission, up to 7 days
  As measured by medical record review (Pre-implementation)
Proportion of patients who receive palliative care consults | Hospital admission, up to 7 days
  As measured by medical record review (Post-implementation)
Proportion of patients who are discharged to hospice | Hospital discharge, up to 7 days
  As measured by medical record review (Pre-implementation)
Proportion of patients who are discharged to hospice | Hospital discharge, up to 7 days
  As measured by medical record review (Post-implementation)
Proportion of patients who have an appointment to the palliative care clinic | Up to 1 month
  As measured by medical record review (Pre-implementation)
Proportion of patients who have an appointment to the palliative care clinic | Up to 1 month
  As measured by medical record review (Post-implementation)

CONTACTS AND LOCATIONS:
Overall Officials: Sendak Mark, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No